CLINICAL TRIAL: NCT01866891
Title: Effects of Regular Perdialytic Physical Activity on the Peripheral Microcirculation in Chronic Hemodialysis Patients
Brief Title: Effects of Physical Activity on the Microcirculation in Hemodialysis Patients
Acronym: ACTIVDIAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012.744
Record Dates: First submitted 2013-05-22; First posted 2013-06-03 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Hemodialysis Patients
Keywords: hemodialysis; microcirculation; physical perdialytic activity; cycling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single arm (Experimental)
  Interventions: Other: Three months of regular perdialytic physical activity (cycling)

INTERVENTIONS:
Other: Three months of regular perdialytic physical activity (cycling) — Cycling, in lying position, at a rate of thirty minutes per dialysis session (three a week), regardless of performance

SUMMARY:
Chronic kidney disease (CKD) is associated with high level of peripheral arterial disease (PAD). This could lead wounds, infections then amputations or deaths by impairment of the peripheral cutaneous perfusion. Medical therapies are presently unable to cure, but only slow down these disorders. Impact of exercise and lower extremity PAD rehabilitation is decreased by the significant inactivity of the chronic hemodialysis patients. Recently, many studies have shown several various favorable effects of the perdialytic physical activity. There is currently no data about effects of the perdialytic activity on the lower extremity perfusion. The aim of this clinical study is to show the impact of three months perdialytic cycling on the microcirculation, in chronic hemodialysis patients. Primary outcome will be the increase of cutaneous perfusion, assessed by measuring transcutaneous oxygen pressure (tcPO2) on about twenty patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients performing chronic hemodialysis for more than 3 months
* Adult aged > or = 18 years old
* Information letter delivered to subjects
* Written free informed consent
* Clinically stable patients
* Voluntary patients to perform 30 minutes cycling per dialysis session
* Social French Security Affiliated subjects

Exclusion Criteria:

* Subjects without inclusion criteria
* Pregnant women
* Subjects protected by the law
* Physical impossibility to achieve exercise
* Medical contraindication to perform physical exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Increase of cutaneous lower extremity perfusion. | TcPO2 will be performed at the inclusion and just after the end of the three month study period

SECONDARY OUTCOMES:
Vascular assessment : Doppler and Index of systolic blood pressure | At the inclusion and after the end of the three month study period
Related quality of life | at the inclusion and after the end of the three month study period
Appetite (score) | at the inclusion and after the end of the three month study period
Daily activity (Seven days pedometers) | at the inclusion and after the end of the three month study period
Protein intake (n-PCR) | at the inclusion and after the end of the three month study period
nutritional biological status (creatinin, albumin and transthyretin protein level) | at the inclusion and after the end of the three month study period
strength (handgrip test) | at the inclusion and after the end of the three month study period

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Edouard Herriot, Lyon, France

REFERENCES:
- [Result] Pelletier C., Jolivot A., Kalbacher E., Long A., Juillard L. Impact de la pratique d'une activité physique régulière perdialytique sur la microcirculation des membres inférieurs chez les patients hémodialysés chroniques : résultats de l'étude Activdial. Néphrologie & Thérapeutique. 2015;11(5):263. doi:10.1016/j.nephro.2015.07.015.
- [Result] Panaye, M., Jolivot, A., Lemoine, S., Villar, E., Fouque, D., & Laville, M. (2014). Outcome and prognosis factors of pregnancies in hemodialysis patients. Nephrology Dialysis Transplantation, 29(Suppl 3), iii520. Poster presented at the 51st ERA-EDTA Congress, Amsterdam, Netherlands.